CLINICAL TRIAL: NCT05872347
Title: A Phase II Study of SPH4336 in Combination With Endocrine Therapy in HR-positive, HER2-negative Breast Cancer Patients With Brain Metastases.
Brief Title: Efficacy and Safety of SPH4336 in Combination With Endocrine Therapy in Breast Cancer Patients With Brain Metastases.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH4336-202
Record Dates: First submitted 2023-05-14; First posted 2023-05-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Brain Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPH4336 Tablets (Experimental): SPH4336 Tablets; Letrozole tablets; Fulvestrant; Exemestane
  Interventions: Drug: SPH4336 Tablets

INTERVENTIONS:
Drug: SPH4336 Tablets — SPH4336 Tablets ：Administered by oral; Letrozole tablets：Administered by oral; Fulvestrant injection：Administered by intravenous infusion; Exemestane：Administered by oral.

SUMMARY:
This study evaluated the safety and efficacy of SPH4336 in combination with endocrine therapy in breast cancer Patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate in this study, completely understand this study, and voluntarily sign the informed consent form (ICF).
2. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 or 1.
3. Life expectancy ≥ 3 months.
4. Patients with locally advanced or metastatic breast cancer who are unable to receive radical surgeries/other local therapies.
5. At least one measurable lesion .
6. Laboratory test results meet the relevant requirements for organ function.
7. Subjects who agree to take effective contraceptive measures.

Exclusion Criteria:

1. Inflammatory breast cancer.
2. Patients unsuitable for endocrine therapy at the investigator's discretion.
3. Have a History of other malignancies prior to the start of study treatment.
4. Taking anti-tumor traditional Chinese patent medicines at the time of signing the ICF.
5. Patients who underwent a surgery prior to the start of study treatment, and have not yet recovered from adverse reactions of the surgery.
6. Patients who participated in a clinical trial and received other investigational drugs before the start of study treatment.
7. Pregnant or lactating women.
8. History of myocardial infarction, unstable angina pectoris, severe arrhythmia, and symptomatic congestive heart failure before the start of study treatment; ≥ NYHA (New York Heart Association) Class II; QTcF≥ 470 ms; left ventricular ejection fraction ≤ 50%.
9. History of ischemic stroke or severe thromboembolic disease before the start of study treatment.
10. Hepatitis B surface antigen positive and HBV (Hepatitis B Virus) DNA > 2,000 IU/mL or > 10(4) copies/mL; HCV (Hepatitis C Virus) antibody positive and HCV RNA positive; or known HIV infection.
11. History of severe allergic diseases, history of severe drug allergies, or known allergy to any ingredient of the investigational product.
12. Presence of diseases or conditions that may impact drug administration or gastrointestinal absorption before the start of study treatment.
13. Presence of uncontrolled infections before the start of study treatment.
14. Known history of drug abuse, excessive drinking, or illegal drug use; history of confirmed neurological or mental disorders.
15. Presence of other diseases that the risks of receiving the study treatment outweigh its benefits, as determined by the investigator, or any other reason for which patients are ineligible for the study as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 52 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial Objective response rate（iORR） | Approximately 3 years
  Objective response rate according to response assessment in neuro-oncology-brain metastases (RANO-BM) criteria.

SECONDARY OUTCOMES:
Intracranial Duration of remission (iDOR) | Approximately 3 years
  DoR is measured from the date of first evidence of a confirmed response (CR or PR), as defined by RANO-BM, to the date objective progression or death from any cause.
Intracranial Disease control rate (iDCR) | Approximately 3 years
  Percentage of participants with BOIR of CR, PR, or SD: IDCR, as defined by RANO-BM is reported.
Progression-free survival (PFS) | Approximately 3 years
  measured by RANO-BM and RECIST 1.1
Overall Survival (OS) | Approximately 8 years
  Determination of the overall survival times of all patients.
Extracranial Objective response rate（eORR） | Approximately 3 years
  Objective response rate according to response assessment in neuro-oncology-brain metastases (RANO-BM) criteria.
Extracranial Disease control rate (eDCR) | Approximately 3 years
  Percentage of participants with BOIR of CR, PR, or SD: IDCR, as defined by RANO-BM is reported.
Extracranial Duration of remission (eDOR) | Approximately 3 years
  DoR is measured from the date of first evidence of a confirmed response (CR or PR), as defined by RANO-BM, to the date objective progression or death from any cause.
Cmax | Approximately 3 years
  PK (Pharmacokinetics) parameters
Tmax | Approximately 3 years
  PK (Pharmacokinetics) parameters
Safety and tolerability | Approximately 3 years
  Adverse event type, incidence, correlation with study drug

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Anhui provincial hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Affiliated Cancer Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Liuzhou people's Hospital, Liuchow, Guangxi
  - Anyang Cancer Hospital, Anyang, He'nan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, He'nan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University cancer Hospital, Harbin, Heilongjiang
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The second people's hospital of neijiang, Neijiang, Sichuan
  - Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang cancer Hospital, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Chongqing University Three Gorges Hospital, Chongqing
  - Guangxi Medical University Cancer Hospital & Guangxi Cancer Institute, Nanning
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Xi'An International Medical Cancer Hospital, Xi'an
  - Henan Cancer Hospital, Zhengzhou